CLINICAL TRIAL: NCT07257432
Title: a Spilt Mouth Clinical Comparative Evaluation of the Electronic Anesthetic Efficacy
Brief Title: Electronic Anesthetic Efficacy Prof. Ali Rokia Ph.D. Al-Andalus University Prof . Mouetaz Kheirallah Ph.D ArabUST
Acronym: ArabUST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mouetaz Kheirallah (Other)
Responsible Party: Sponsor-Investigator, Mouetaz Kheirallah, Ph.D., OMFS, DDS, Associate Professor, Arab University for Science and Technology
Organization: Arab University for Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ArabUST
Record Dates: First submitted 2025-11-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pain Perception
Keywords: Dental Anesthesia

STUDY DESIGN:
Intervention Model Description: The split-mouth design was applied to the study group, with one arm for therapeutic intervention involving Smartject injection , and the other arm involving traditional injectors
Who Masked: Care Provider, Investigator
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic syringe therapeutic intervention arm (Experimental): During the appointment, the subjects randomly received 1.8 ml of 2% plain lidocaine for the Intraoral Mental nerve block on both sides (experimental and control). A Carpule syringe with an aspiration and short needles 30G were used on the control side, while Smartject was used on the experimental side
  Interventions: Drug: Experimental group: Electronic syringe therapeutic intervention arm; Drug: control group: therapeutic intervention using a traditional syringe
- therapeutic intervention using a traditional syringe (Experimental): During the appointment, the subjects randomly received 1.8 ml of 2% plain lidocaine for the Intraoral Mental nerve block on both sides (experimental and control). A Carpule syringe with an aspiration and short needles 30G were used on the control side, while Smartject was used on the experimental side
  Interventions: Drug: Experimental group: Electronic syringe therapeutic intervention arm; Drug: control group: therapeutic intervention using a traditional syringe

INTERVENTIONS:
Drug: Experimental group: Electronic syringe therapeutic intervention arm — Intraoral Mental nerve block on both sides (experimental and control). A Carpule syringe with an aspiration and short needles 30G were used on the control side, while Smartject was used on the experimental side
  Other Names: anesthesia pen x
Drug: control group: therapeutic intervention using a traditional syringe — During the appointment, the subjects randomly received 1.8 ml of 2% plain lidocaine for the Intraoral Mental nerve block on both sides (experimental and control). A Carpule syringe with an aspiration and short needles 30G were used on the control side
  Other Names: surgimax

SUMMARY:
A Spilt Mouth Clinical Comparative Evaluation Of The Electronic Anesthetic Efficacy Comparison of traditional local anesthesia with electronic local anesthesia in terms of the ability to reduce pain during injection and the duration of the anesthetic effect

DETAILED DESCRIPTION:
Study Design:

The mouth will be split in half using a split mouth study. The lower anterior teeth will be injected with a conventional local anesthetic syringe on one side, and the patient will be injected with an electronic anesthetic syringe on the other side.

The study will be conducted on a sample of volunteers aged 18 to 30 years at the Faculty of Dentistry at Al-Andalus University.

The objectives and procedure will be explained to each group of patients, and informed consent will be obtained from each patient to accept the research procedures.

A 2% non-vasoconstrictor lidocaine local anesthetic will be used for all patients.

ELIGIBILITY:
Inclusion Criteria:". Age ranged from 20 to 30 years , no menstrual cycle, The participants were not allergic to local anesthetics, had not used medication that would alter pain perception, none of them had not ever experienced Smartject injection before, and none of them were alcoholics or smokers, The participants were not allergic to local anesthetics.

Exclusion Criteria:

allergic to local anesthetics ,females during menstural cycle ,bad oral care.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Onset time | 2 month
  was considered as the period between the end of the injection and the first subsequent Onset time was considered as the period between the end of the injection and the first subsequent readings without response. After this period, the tooth was tested every 10 minutes until readings returned to the baseline threshold. Each subject was asked to record the time of return to normal sensation in the lower lip

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 month
  VAS uses a straight horizontal line of extent measuring 10 cm. The ends state the maximum limit of pain orientated from the best (right) to the worst (left) so that the patient can indicate the intensity of the pain (0-100). The intensity of pain is made by measuring the dimension from "no pain" to "very severe pain" based on the patient's signs

OTHER OUTCOMES:
duration of the anesthesia | 2 month
  was asked to record the time of return to normal sensation in the lower lip

CONTACTS AND LOCATIONS:
Overall Officials: Ali G Rokia, ph.D, Study Chair — Al-Andalus University
Locations (2):
- Syria (2):
  - Al Andalus University, Tartus, Al Kadmous
  - Arab University, Hama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Douglas BL. Electronic dental anesthesia. Anesth Prog. 1993;40(3):99-100. No abstract available. PMID 7645794